CLINICAL TRIAL: NCT00311155
Title: Treat-to-Target Study of Olmesartan Medoxomil and an Add-on Treatment Algorithm Consisting of Hydrochlorothiazide and Amlodipine Besylate in Patients With Mild to Moderate Hypertension
Brief Title: Olmesartan and an add-on Treatment in Patients With Mild to Moderate Hypertension
Acronym: OLMETREAT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sankyo Pharma Gmbh (Industry)
Responsible Party: Senior Manager - Study Coordination, Daiichi Sankyo Europe, GmbH
Organization: Daiichi Sankyo (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SP-OLM-03-05; 2005-004659-36 (EudraCT Number)
Record Dates: First submitted 2006-04-03; First posted 2006-04-05 (Estimated); Results first posted 2010-11-10 (Estimated); Last update posted 2010-12-10 (Estimated); Status verified 2010-11

CONDITIONS: Essential Hypertension
Keywords: Olmesartan medoxomil; Hypertension
MeSH Terms: conditions — Essential Hypertension; Hypertension | interventions — Olmesartan Medoxomil; Hydrochlorothiazide; Amlodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Olmesartan medoxomil oral tablets for 4 weeks followed by, if necessary:
  Olmesartan medoxomil oral tablets + hydrochlorothiazide oral tablets for 8 weeks, followed by, if necessary:
  Olmesartan medoxomil oral tablets + hydrochlorothiazide oral tablets + amlodipine oral tablets for 8 weeks
  Interventions: Drug: olmesartan medoxomil + hydrochlorothiazide, if necessary + amlodipine, if necessary

INTERVENTIONS:
Drug: olmesartan medoxomil + hydrochlorothiazide, if necessary + amlodipine, if necessary — Olmesartan medoxomil oral tablets 20 mg for 4 weeks followed by, if necessary: Olmesartan medoxomil oral tablets 20 mg + hydrochlorothiazide oral tablets 12.5 mg for 4 weeks, followed by, if necessary: Olmesartan medoxomil oral tablets 20 mg + hydrochlorothiazide oral tablets 25 mg for 4 weeks, followed by, if necessary: Olmesartan medoxomil oral tablets 20 mg + hydrochlorothiazide oral tablets 25 mg + amlodipine oral tablets 5 mg for 4 weeks, followed by, if necessary: Olmesartan medoxomil oral tablets 20 mg + hydrochlorothiazide oral tablets 25 mg + amlodipine oral tablets 10 mg for 4 weeks. All study medications are to be taken once daily. The subject's participation completes when blood pressure goals are achieved.

SUMMARY:
This study is to assess the safety and efficacy of an add-on treatment algorithm with olmesartan, hydrochlorothiazide and amlodipine in patients with mild to moderate hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients age greater than or equal to 18 years with mild to moderate hypertension.
* Pre-treated patients with normal or elevated blood pressure (BP) are eligible to participate if their pre-treatment medication can be withdrawn. At the end of the placebo run-in period sitting systolic BP greater than or equal to 140 and less than 180 mmHg and/or sitting diastolic BP greater than or equal to 90 and less than 110 mmHg at trough.

Exclusion Criteria:

* Female patients of childbearing potential must not be pregnant or lactating and must be using adequate contraception.
* Patients with serious disorders which may limit the ability to evaluate the efficacy or safety of the test drug(s), including cardiovascular, renal, pulmonary, hepatic, gastrointestinal, endocrine/metabolic, haematological/oncological, neurological and psychiatric diseases.
* Patients within the last 6 months having a history of myocardial infarction, unstable angina pectoris, percutaneous coronary intervention, heart failure, cerebrovascular accident, or transient ischemic attack.
* Patients with clinically significant elevations in laboratory values at Screening Visit.
* Patients with secondary hypertension of any etiology, such as renal disease, pheochromocytoma, or Cushing's syndrome.
* Patients with contraindications for olmesartan medoxomil, hydrochlorothiazide, and/or amlodipine besylate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 694 (Actual)
Dates: Start 2006-03; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Heagerty, MD, Principal Investigator — University of Manchester, Dept. of Medicine
Locations (79):
- Austria (6):
  - Fulpmes
  - University Klinik, F. Innere Medizin, Innsbruck
  - Innsbruck
  - Kundl
  - Salzburg
  - Diakonissen-Krankenhaus Hospital, Salzburg-Aigen
- Belgium (4):
  - Brussels
  - Mechelen
  - Centre Hospitalier du Bois de l'Abbaye et de Hesba, Department of Intensive Care, Seraing
  - Allgemeen Ziekenhuis Maria-Middelares, Cardiologie, Campus de Pelikaan, Temse
- France (14):
  - Ancerville
  - Bourges
  - Derval
  - Grenoble
  - Lille
  - Montrevel-en-Bresse
  - Pouilly-en-Auxois
  - Poussan
  - Saint-Aubin-des-Châteaux
  - Saint-Étienne-de-Montluc
  - Saint-Priest
  - Sorcy-Saint-Martin
  - Strasbourg
  - Yerres
- Germany (14):
  - Annweiler am Trifels
  - Balve
  - Bammental
  - Ev. Krankenhaus Bielefeld, Medizinische Klinik in Bethel - Gilead I, Bielefeld
  - Uniklinik Bonn, Bonn
  - Goch
  - Haag
  - Hamburg
  - Heidelberg
  - Heidelberg (Neuenheim)
  - Mühldorf / Inn
  - Schwenningen
  - VS-Villingen
  - Weyhe
- Italy (13):
  - Ospedale Regina Apostolorum, Albano Laziale (RM)
  - Ospedale C.G. Mazzoni, Ascoli Piceno
  - Ospedale Nuovo Cutroni, Barcellona Pozzo Di Gotto (ME)
  - Casa di Cura "La Madonnina", Bari
  - Ospedale San Sebastiano, Caserta
  - Ospedale Vittorio Emanuele, Catania
  - Università degli Studi "G. D'Annunzio", Chieti Scalo
  - Azienda Ospedaliera "Madonna delle Grazie", Matera
  - Ospedale San Paolo, Milan
  - Ospedale San Carlo Borromeo, Milan
  - Presidio Ospedaliero San Lorenzo, Palermo
  - Presidio Ospedaliero di Portogruaro, Portogruaro (VE)
  - Azienda Policlinico Universitario a Gestione Diret, Udine
- Netherlands (6):
  - 's-Hertogenbosch
  - Maxima Medisch Centrum, Eindhoven
  - H. Elvas, Elvas
  - Hilversum
  - Lieshout
  - Waalwijk
- Portugal (3):
  - H. Almada, Almada Almada
  - Hospital Fernando da Fonseca, Amadora Amadora
  - Hospital de. S. Marta, Lisboa Lisboa
- Switzerland (5):
  - Zentrum Oberdorf, Affoltern am Albis
  - Bellinzona
  - Gland
  - Petit Lancy
  - Praxis Dreispitz, Zurich
- United Kingdom (14):
  - The Atherstone Surgery, Atherstone
  - The Medical Centre, Birmingham
  - Waterloo Medical Centre, Blackpool
  - Rowden Surgery, Chippenham
  - The Gables Medical Centre, Coventry
  - Bridge Medical Centre, Crawley
  - Homefield Surgery, Exeter
  - Woodside Health Centre, Glasgow
  - Castle Milk Health Centre, Glasgow
  - Division of Cardiovascular and Endocrine Sciences, Manchester
  - University of Manchester, Manchester
  - Oakside Surgery, Plymouth
  - Norwood Medical Centre, Sheffield
  - Lovemead Group Practice, Trowbridge

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted between April 2006 and April 2008 in 9 European countries at 58 investigational sites. The countries participating were: Austria, Belgium, France, Germany, Italy, The Netherlands, Portugal, Switzerland, and United Kingdom.
Groups:
- Olmesartan+Hydrochlorothiazide,if Needed+Amlodipine, if Needed: Olemesartan 20 mg to start. Hydrochlorothiazide 12.5 mg and then 25 mg was added, if necessary. If blood pressure goal was still not achieved, amlodipine 5 mg and then 10 mg were added, if needed. Thus, the maximum combination was olmesartan 20mg + hydrochlorothiazide 25mg + amlodipine 10mg.
Period: Overall Study
Arm/Group | Olmesartan+Hydrochlorothiazide,if Needed+Amlodipine, if Needed
Started | 694
Completed | 601 (Some participants had multiple reasons for discontinuation)
Not Completed | 93
Not completed — Adverse Event | 21
Not completed — Withdrawal by Subject | 17
Not completed — Did not meet entry criteria | 55

BASELINE CHARACTERISTICS:
Arm/Group | Olmesartan+Hydrochlorothiazide,if Needed+Amlodipine, if Needed
Number analyzed (Participants) | 694
Age Continuous [Mean (Standard Deviation); unit: years] | 58.16 (12.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 337
  Male | 357
Region of Enrollment [Number; unit: participants]
  Portugal | 12
  France | 121
  Belgium | 94
  Austria | 35
  Netherlands | 43
  Germany | 207
  United Kingdom | 141
  Italy | 35
  Switzerland | 6
Weight [Mean (Standard Deviation); unit: kg] | 82.16 (16.09)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 28.86 (4.69)
Ethnicity [Number; unit: Participants]
  Caucasian | 678
  Black | 13
  Asian | 3

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Participants Treated to Target Blood Pressure Goals Overall and for Each Treatment Step From Baseline to Completion of Treatment During Which the Goal Was Achieved.
Description: For non-diabetic participants the target seated blood pressure goals were: Systolic - ≤130 mm Hg; Diastolic - ≤85 mm Hg. For diabetic participants the target seated blood pressure goals were: Systolic - <130 mm Hg; Diastolic - <80 mm Hg.
Time Frame: Baseline to ≤20 weeks
Population: 691 = the full analysis set (FAS). FAS consists of all participants who received trial medication and who had data from at least one post-baseline visit with regard to the primary efficacy parameter, i.e., both the systolic and the diastolic blood pressure (BP) had to be measured. N is reduced for each treatment as subjects attain BP goals.
Measure: Number; unit: Percentage of participants
Groups:
- Olmesartan+Hydrochlorothiazide,if Needed+Amlodipine, if Needed: Olmesartan (OLM) 20 mg to start for 4 weeks. Hydrochlorothiazide (HCTZ) 12.5 mg is added, if necessary, for 4 additional weeks. Hydrochlorothiazide is doubled (25 mg), if necessary, for 4 additional weeks. If blood pressure goals were still not achieved, amlodipine (AML) 5 mg was added to the olmesartan and hydroclorothiazide for an additional 4 weeks. Finally, the amplodine was doubled (10 mg), if needed, for the final 4 weeks of treatment. Thus, the maximum combination was olmesartan 20mg + hydrochlorothiazide 25mg + amlodipine 10mg. The subject's participation in the study was concluded as soon as blood pressure goals were met.
Arm/Group | Olmesartan+Hydrochlorothiazide,if Needed+Amlodipine, if Needed
Number analyzed (Participants) | 691
Percentage of participants
  Overall N=691 | 71.8
  OLM 20 mg N=688 | 12.3
  OLM 20 mg+HCTZ 12.5 mg N=580 | 16.4
  OLM 20 mg+HCTZ 25 mg N=446 | 19.2
  OLM 20 mg+HCTZ 25 mg+AML 5 mg N=296 | 14.9
  OLM 20 mg+HCTZ 25 mg+AML 10 mg N=176 | 8.5

2. Secondary Outcome: Percentage of Participants Who Achieved Normalized Blood Pressure Overall and for Each Treatment From Baseline to Completion of the Treatment During Which Blood Pressure Goals Were Achieved
Description: Normalized blood pressure is defined as a mean sitting systolic blood (sBP) pressure at trough of <140 mmHg and mean sitting diastolic blood pressure (dBP)of <90 mmHg for non-diabetic patients or a mean sitting sBP at trough of <130 mmHg and mean sitting dBP <80 mmHg for diabetic patients.
Time Frame: Baseline to ≤20 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Olmesartan+Hydrochlorothiazide,if Needed+Amlodipine, if Needed
Number analyzed (Participants) | 691
Percentage of participants
  Overall N=691 | 84.5
  OLM 20 mg N=688 | 22.7
  OLM 20 mg + HCTZ 12.5 mg N=580 | 31.1
  OLM 20 mg + HCTZ 25 mg N=446 | 32.7
  OLM 20 mg + HCTZ 25 mg + AML 5 mg N=296 | 23.9
  OLM 20 mg + HCTZ 25 mg + AML 10 mg N=176 | 14.8

3. Secondary Outcome: Percentage of Participants Who Were Diastolic Responders Overall and for Each Treatment From Baseline to the Completion of Treatment During Which Blood Pressure Goals Were Achieved.
Description: Diastolic responders were defined as a participant who is a normaliser or has a lowering of the mean sitting diastolic blood pressure of ≥10 mmHg at trough.
Time Frame: Baseline to ≤20 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Olmesartan+Hydrochlorothiazide,if Needed+Amlodipine, if Needed
Number analyzed (Participants) | 691
Percentage of participants
  Overall N=691 | 93.3
  OLM 20 mg N=688 | 36.6
  OLM 20 mg + HCTZ 12.5 mg N=580 | 52.4
  OLM 20 mg + HCTZ 25 mg N=446 | 48.6
  OLM 20 mg + HCTZ 25 mg + AML 5 mg N=296 | 33.4
  OLM 20 mg + HCTZ 25 mg + AML 10 mg N=176 | 20.4

4. Secondary Outcome: Percentage of Participants Who Were Systolic Responders Overall and for Each Treatment From Baseline to the Completion of the Treatment During Which Blood Pressure Goals Were Achieved
Description: Systolic responders defined as a participant who is a normaliser or has a lowering of the mean sitting systolic blood pressure of ≥20 mmHg at trough
Time Frame: Baseline to ≤20 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Olmesartan+Hydrochlorothiazide,if Needed+Amlodipine, if Needed
Number analyzed (Participants) | 691
Percentage of Participants
  Overall N=691 | 92.6
  OLM 20 mg N=688 | 34.2
  OLM 20 mg + HCTZ 12.5 mg N=580 | 49.6
  OLM 20 mg + HCTZ 25 mg N=446 | 46.6
  OLM 20 mg + HCTZ 25 mg + AML 5 mg N=296 | 33.3
  OLM 20 mg + HCTZ 25 mg + AML 10 mg N=176 | 20.5

5. Secondary Outcome: Mean Change in Diastolic Blood Pressure Overall and for Each Treatment From Baseline to the Completion of the Treatment
Time Frame: Baseline to ≤20 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Olmesartan+Hydrochlorothiazide,if Needed+Amlodipine, if Needed
Number analyzed (Participants) | 691
mm Hg
  Overall N=691 | -15.73 (7.98)
  OLM 20 mg N=688 | -6.44 (7.53)
  OLM 20 mg + HCTZ 12.5 mg N=580 | -10.15 (7.54)
  OLM 20 mg + HCTZ 25 mg N=446 | -13.04 (7.67)
  OLM 20 mg + HCTZ 25 mg + AML 5 mg N=296 | -14.03 (8.27)
  OLM 20 mg + HCTZ 25 mg + AML 10 mg N=176 | -14.47 (8.86)

6. Secondary Outcome: Mean Change in Systolic Blood Pressure Overall and for Each Treatment From Baseline to the Completion of the Treatment
Time Frame: Baseline to ≤20 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Olmesartan+Hydrochlorothiazide,if Needed+Amlodipine, if Needed
Number analyzed (Participants) | 691
mm Hg
  Overall N=691 | -29.58 (13.52)
  OLM 20 mg N=688 | -11.97 (11.42)
  OLM 20 mg + HCTZ 12.5 mg N=580 | -19.55 (12.12)
  OLM 20 mg + HCTZ 25 mg N=446 | -24.51 (13.14)
  OLM 20 mg + HCTZ 25 mg + AML 5 mg N=296 | -27.06 (13.72)
  OLM 20 mg + HCTZ 25 mg + AML 10 mg N=176 | -28.02 (13.52)

ADVERSE EVENTS:
Time Frame: The time frame was from baseline to up to 20 weeks of treatment
Description: Safety was addressed in terms of occurrences of adverse envents (AEs), of treatment-emergent AEs, changes in vital signs, ECGs, physical examination findings and laboratory parameters. AEs were documented during the whole study period by spontaneous reports to the investigator or upon questioning by or observations by the investigator.
Arm/Group | Olmesartan+Hydrochlorothiazide,if Needed+Amlodipine, if Needed
Serious Adverse Events (participants affected / at risk) | 7/694
Other Adverse Events (participants affected / at risk) | 293/694
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Olmesartan+Hydrochlorothiazide,if Needed+Amlodipine, if Needed (N=694)
Renal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cellulitis (Infections and infestations) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Myocardial infacrtion (Cardiac disorders) | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Olmesartan+Hydrochlorothiazide,if Needed+Amlodipine, if Needed (N=694)
bronchitis (Infections and infestations) | 46
Urinary tract infection (Infections and infestations) | 26
Nasopharyngitis (Infections and infestations) | 17
Upper respiratory tract infection (Infections and infestations) | 17
Dizziness (Nervous system disorders) | 77
Headache (Nervous system disorders) | 23
cough (Respiratory, thoracic and mediastinal disorders) | 15
Back pain (Musculoskeletal and connective tissue disorders) | 25
Pain in extremity (Musculoskeletal and connective tissue disorders) | 15
Oedema peripheral (General disorders) | 32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No